CLINICAL TRIAL: NCT00376766
Title: Rapid Oral Treatment of Cluster Epileptic Seizures. Efficacy Assessment of Levetiracetam in Cluster Seizures.
Brief Title: Clinical Trial : TROCC (Quick Oral Treatment of Cluster Epileptic Seizures)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment recruitment recruitment recruitment difficulties
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DTCIC 05 24
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Epilepsy; Drug Resistant
Keywords: Cluster seizure; seizure clustering; repetitive seizure; Drug resistant epilepsy; Levetiracetam; keppra
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: levetiracetam

SUMMARY:
This is a double blind, placebo controlled, add-on clinical trial, of levetiracetam efficacy and safety, in epilepsy cluster seizure.

Efficacy is evaluated in the range of 2 to 24 hours after taking the tablet. If the patient has a seizure during this interval, he is considered as a non-respondent patient.

DETAILED DESCRIPTION:
Seizure clustering has been defined as a series of unusual frequency of seizures with return to baseline between events. The most common definition of cluster seizure is three seizures per 24 hours.

The usual treatment of cluster seizure is benzodiazepin. This is recognized efficient therapy but has many side effects. Thus it is important to develop as an new therapeutic to improve patient care. Levetiracetam is an antiepileptic drug used in addition to other antiepileptic drugs with less side effects than benzodiazepin.

The aim of this study is to evaluate the effectiveness and safety of levetiracetam in epilepsy cluster seizure.

This is a double blind, placebo controlled, add-on clinical trial with two phases :

Phase 1 : Double blind phase during 24 hours (H0 to H24). After consent signature and randomization, the patient takes two tablets of levetiracetam or placebo. If the patient has a seizure between H3 and H24, he is considered as a non-respondent patient. If there is a risk of rapid evolution to an statue epilepticus, the investigator can break the blind and adapt the patient treatment accordingly.

Phase 2 : This is an open phase after H24. this phase consists of breaking the blind with free adaption of the therapy by the investigator, and patients follow-up during 1 month.

The randomization is stratify by center. The size of randomization blocks is random because of the systematic breaking blind after 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65
* Drug resistant epilepsy, partial seizure
* Epilepsy diagnosed for more than 2 years
* Epilepsy treated for more than 1 year with no change of treatment in the month before the enrolment
* Onset of cluster seizure in the 24 hours before enrolment
* For women : effective contraception
* Affiliation to the French social security

Exclusion Criteria:

* Inability to tolerate levetiracetam, likely poor compliance
* Patient taking antiepileptic treatment (benzodiazepine) in addition to current treatment during the last 48h00.
* Patient taking 1g/day of levetiracetam with Creatinin clearance < 50ml/min
* Patient taking 2g/day of levetiracetam with Creatinin clearance < 80ml/min
* Patient taking more than 2g/day of levetiracetam
* Hepatic or cardiovascular pathology
* Progressive psychiatric pathology
* Degenerative neurologic disease
* Cluster seizure due to an acute symptomatic reason
* Disorder of consciousness
* Suspicion of status epilepticus or rapid evolution to status epilepticus
* Suspicion of psychogenic nonepileptic seizure
* Pregnant woman or nursing woman
* Suicidal thoughts
* Incapacity to give consent, minor patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Ratio of patients who are free of seizure between H3 and H24 in both groups.

SECONDARY OUTCOMES:
Items 1,2,3 of the Clinical Global Impression scale.
Side effects during the study.
Time between H0 and the last seizure.
Type and ratio of epileptic fit between H0 and H24.
Number of seizures occured between H3 and H10, H10 and H17, H17 and H24, corresponding to the half-time of the treatment (7 hours).
Description of therapeutic adaptation at 1 month after patient enrolment.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Maillard, Dr, Principal Investigator — Central Hospital, Nancy, France; Serge CHASSAGNON, Dr, Principal Investigator — University Hospital of Strasbourg; Cecile SABOURY, Dr, Principal Investigator — University Hospital of Strasbourg; Edouard HIRSH, Dr, Principal Investigator — University Hospital of Strasbourg; William SZHURAJ, Dr, Principal Investigator — University Hospital of Lille; Philippe DERAMBURE, Dr, Principal Investigator — University Hospital of Lille; Jerome PETIT, Dr, Principal Investigator — La Teppe Institution; Vincent TAREL, Dr, Principal Investigator — Regional Hospital of Chambery; Dominique ROSENBERG, Dr, Principal Investigator — University Hospital, Clermont-Ferrand; Helene CATENOIX, Dr, Principal Investigator — University Hospital of Lyon; Philippe RYVELIN, Dr, Principal Investigator — University Hospital of Lyon; Philippe CONVERS, Dr, Principal Investigator — University Hospital of St Etienne; Pierre THOMAS, Dr, Principal Investigator — University Hospital of Nice
Locations (10):
- France (10):
  - Neurology department, Nice, Alpes de Haute provence
  - Etablissement la Teppe, Tain-l'Hermitage, Drome
  - Neurology department, Grenoble, Isere
  - Neurology department, Lille, Nord
  - Neurology department, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - Neurology department, Clermont-Ferrand, Puy de Dome
  - Neurology department, Lyon, Rhone
  - Neurology Department, Chambéry, Savoie
  - Neurology department, Nancy
  - Neurology department, Strasbourg

REFERENCES:
- [Background] Haut SR, Shinnar S, Moshe SL. Seizure clustering: risks and outcomes. Epilepsia. 2005 Jan;46(1):146-9. doi: 10.1111/j.0013-9580.2005.29004.x. PMID 15660781
- [Background] Dreifuss FE, Rosman NP, Cloyd JC, Pellock JM, Kuzniecky RI, Lo WD, Matsuo F, Sharp GB, Conry JA, Bergen DC, Bell WE. A comparison of rectal diazepam gel and placebo for acute repetitive seizures. N Engl J Med. 1998 Jun 25;338(26):1869-75. doi: 10.1056/NEJM199806253382602. PMID 9637805
- [Background] Mitchell WG, Conry JA, Crumrine PK, Kriel RL, Cereghino JJ, Groves L, Rosenfeld WE. An open-label study of repeated use of diazepam rectal gel (Diastat) for episodes of acute breakthrough seizures and clusters: safety, efficacy, and tolerance. North American Diastat Group. Epilepsia. 1999 Nov;40(11):1610-7. doi: 10.1111/j.1528-1157.1999.tb02047.x. PMID 10565590
- [Background] Shorvon SD, Lowenthal A, Janz D, Bielen E, Loiseau P. Multicenter double-blind, randomized, placebo-controlled trial of levetiracetam as add-on therapy in patients with refractory partial seizures. European Levetiracetam Study Group. Epilepsia. 2000 Sep;41(9):1179-86. doi: 10.1111/j.1528-1157.2000.tb00323.x. PMID 10999557
- [Background] Cereghino JJ, Biton V, Abou-Khalil B, Dreifuss F, Gauer LJ, Leppik I. Levetiracetam for partial seizures: results of a double-blind, randomized clinical trial. Neurology. 2000 Jul 25;55(2):236-42. doi: 10.1212/wnl.55.2.236. PMID 10908898